CLINICAL TRIAL: NCT06632951
Title: A Phase 2, Open-Label, Randomized Study of Livmoniplimab in Combination With Budigalimab Versus Chemotherapy in Subjects With Metastatic Urothelial Carcinoma
Brief Title: Study to Evaluate Adverse Events and Change in Disease Activity When Intravenously (IV) Infused Livmoniplimab is Used in Combination With IV Infused Budigalimab in Adult Participants With Urothelial Carcinoma (UC)
Acronym: LIVIGNO-3
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M25-204; 2024-515506-11-00 (Other: EU CT)
Record Dates: First submitted 2024-10-08; First posted 2024-10-09 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Urothelial Carcinoma
Keywords: Urothelial Carcinoma; Metastatic Urothelial Carcinoma; Docetaxel; Paclitaxel; Gemcitabine; Livmoniplimab; Budigalimab; ABBV-181; ABBV-151; Cancer; LIVIGNO-3
MeSH Terms: conditions — Carcinoma, Transitional Cell; Neoplasms | interventions — budigalimab; Docetaxel; Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: Livmoniplimab (Dose A) + Budigalimab (Experimental): Participants will receive livmoniplimab (dose A) in combination with budigalimab, as part of the approximately 3.5 years study duration.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Arm 2: Livmoniplimab (Dose B) + Budigalimab (Experimental): Participants will receive livmoniplimab (dose B) in combination with budigalimab, as part of the approximately 3.5 years study duration.
  Interventions: Drug: Livmoniplimab; Drug: Budigalimab
- Arm 3: Docetaxel, Paclitaxel, or Gemcitabine (Experimental): Participants will receive docetaxel, paclitaxel, or gemcitabine, investigator's choice, as part of the approximately 3.5 years study duration.
  Interventions: Drug: Docetaxel; Drug: Paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Livmoniplimab — Intravenous (IV) Infusion
  Other Names: ABBV-151
  Arms: Arm 1: Livmoniplimab (Dose A) + Budigalimab; Arm 2: Livmoniplimab (Dose B) + Budigalimab
Drug: Budigalimab — IV Infusion
  Other Names: ABBV-181
  Arms: Arm 1: Livmoniplimab (Dose A) + Budigalimab; Arm 2: Livmoniplimab (Dose B) + Budigalimab
Drug: Docetaxel — IV Infusion
  Arms: Arm 3: Docetaxel, Paclitaxel, or Gemcitabine
Drug: Paclitaxel — IV Injection
  Arms: Arm 3: Docetaxel, Paclitaxel, or Gemcitabine
Drug: Docetaxel — IV Injection
  Arms: Arm 3: Docetaxel, Paclitaxel, or Gemcitabine
Drug: Paclitaxel — IV Infusion
  Arms: Arm 3: Docetaxel, Paclitaxel, or Gemcitabine
Drug: Gemcitabine — IV Infusion
  Arms: Arm 3: Docetaxel, Paclitaxel, or Gemcitabine

SUMMARY:
Urothelial carcinoma (UC) is the ninth most common cancer type worldwide. While the treatment of front-line metastatic urothelial carcinoma (mUC) has improved, there remains a high unmet need for effective therapies for participants who have recurrent disease and disease that has progressed after frontline treatment. The purpose of this study is to evaluate the optimized dose, adverse events, and efficacy of livmoniplimab in combination with budigalimab.

Livmoniplimab is an investigational drug being developed for the treatment of mUC. There are 3 treatment arms in this study and participants will be randomized in a 1:1:1 ratio. Participants will either receive livmoniplimab (at one of 2 different doses) in combination with budigalimab (another investigational drug), or either docetaxel, paclitaxel, or gemcitabine (based on investigator's choice). Approximately 150 adult participants will be enrolled in the study across 56 sites worldwide.

In arm 1, participants will receive intravenously (IV) infused livmoniplimab (dose A) in combination with IV infused budigalimab. In arm 2, participants will receive IV infused livmoniplimab (dose B) in combination with IV infused budigalimab. In arm 3 (control), participants will receive the investigator's choice: IV infused or injected docetaxel; IV infused or injected paclitaxel; or IV infused gemcitabine. The estimated duration of the study is up to approximately 3.5 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, questionnaires, and scans.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically or cytologically confirmed urothelial carcinoma (i.e., cancer of the bladder, renal pelvis, ureter, or urethra). Mixed histologic types are allowed if urothelial (transitional cell) is the predominant histology.
* Participant has radiologically documented metastatic disease.
* Participant must have experienced radiographic progression or relapse on checkpoint inhibitor (anti-programmed cell death protein 1 [PD-1] or anti-programmed death-ligand 1 [PD-L1]) in the metastatic, adjuvant, or neo-adjuvant setting. Participant must have received at least 2 cycles of anti-PD-1 or anti-PD-L1.
* Participants eligible for platinum must have received a platinum containing regimen (cisplatin or carboplatin) in the metastatic, locally advanced, neoadjuvant, or adjuvant setting. If platinum was administered in the neoadjuvant or adjuvant setting, participant must have progressed within 6 months of completion of treatment. Platinum ineligible participants may enroll in this study without receiving a platinum containing regimen.
* Participant has at least 1 measurable lesion per response evaluation criteria in solid tumors (RECIST) v1.1 as determined by investigator.
* Life expectancy must be at least 3 months.

Exclusion Criteria:

* Participant has received more than 1 prior chemotherapy regimen for urothelial cancer in metastatic setting, including chemotherapy agents planned in comparator arm.

  * Platinum based chemotherapy administered in adjuvant or neoadjuvant setting will count towards this criterion if participant progressed within 6 months of completion.
  * Chemotherapy administered during concurrent chemoradiotherapy for primary cancer will not count towards this criterion.
  * The substitution of carboplatin for cisplatin does not constitute a new regimen provided no new chemotherapeutic agents were added to the regimen and no progression was noted prior to the change in platinum.
  * Antibody-drug conjugate (ADC) will not count towards this criterion.
  * Participant who previously received gemcitabine in combination with platinum in metastatic setting will be eligible to receive docetaxel or paclitaxel in comparator arm.
* Participant has received more than 1 antibody-drug conjugate (ADC) in metastatic setting.
* Has had prior radiation therapy within 28 days prior to first dose of study drug or who has not recovered (i.e., <= Grade 1 or at baseline) from adverse events due to radiotherapy.
* History of additional malignancy or history of prior malignancy, except for adequately treated basal or squamous skin cancer, or cervical carcinoma in situ without evidence of disease, or malignancy treated with curative intent and with no evidence of disease recurrence for 5 years since the initiation of that therapy.
* Prior allogeneic stem cell or solid organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to Approximately 3.5 Years
  OS is defined as the time measured from randomization until death from any cause.

SECONDARY OUTCOMES:
Progression-Free survival (PFS) | Up to Approximately 3.5 Years
  PFS is defined as the time measured from randomization until the first documentation of progressive disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as determined by investigators or death from any cause, whichever occurs first.
Best Overall Response (BOR) per Investigator | Up to Approximately 3.5 Years
  BOR is defined as achieving complete response (CR) or partial response (PR) according to RECIST 1.1 as determined by investigators at any time prior to subsequent anticancer therapy.
Duration of Response (DOR) per Investigator | Up to Approximately 3.5 Years
  DOR id defined as the time from first CR/PR until the first documentation of progressive disease according to RECIST 1.1 as determined by investigators or death from any cause, whichever occurs first.
Percentage of Participants with Adverse Events (AE)s | Up to Approximately 3.5 Years
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Percentage of Participants with Serious Adverse Events (SAE)s | Up to Approximately 3.5 Years
  An SAE is defined as an AE that results in the death of the participant, threat to the participant's life, hospitalization, congenital abnormality, persistent or significant disability/incapacitation, or medical event requiring medical or surgical interventions to prevent a serious outcome.
Percentage of Participants with Treatment Emergent Adverse Events (TEAE)s | Up to Approximately 3.5 Years
  The treatment-emergent period is defined as time from the date of the first dose of study drug up to 90 days after the date of the last dose of study drug, or the first date starting new anticancer therapy, whichever occurs earlier. TEAEs include all AEs that occurred or worsened during the treatment emergent period and all treatment related SAEs as assessed by investigators.
Percentage of Participants with Clinically Significant Vital Sign Measurements as Assessed by the Investigator | Up to Approximately 3.5 Years
  Vital signs are defined as systolic and diastolic blood pressure, pulse rate, respiratory rate, and body temperature.
Percentage of Participants with Clinically Significant Laboratory Values | Up to Approximately 3.5 Years
  Percentage of participants with clinically significant laboratory values (hematology, chemistry, coagulation, and urinalysis) as assessed by the investigator.
Percentage of Participants with Immune-Related Reactions as AEs of Special Interest | Up to Approximately 3.5 Years
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Maximum Observed Serum Concentration (Cmax) of Livmoniplimab | Up to Approximately 3.5 Years
  Cmax is defined as the maximum observed serum concentration of livmoniplimab.
Cmax of Budigalimab | Up to Approximately 3.5 Years
  Cmax is defined as the maximum observed serum concentration of budigalimab.
Time to Reach Cmax (Tmax) of Livmoniplimab | Up to Approximately 3.5 Years
  Tmax is defined as the time to reach Cmax of livmoniplimab.
Tmax of Budigalimab | Up to Approximately 3.5 Years
  Tmax is defined as the time to reach Cmax of budigalimab.
Area Under the Serum Concentration Versus Time Curve (AUC) of Livmoniplimab | Up to Approximately 3.5 Years
  AUC is defined as the area under the serum concentration versus time curve of livmoniplimab.
AUC of Budigalimab | Up to Approximately 3.5 Years
  AUC is defined as the area under the serum concentration versus time curve of budigalimab.
Clearance (CL) of Livmoniplimab | Up to Approximately 3.5 Years
  CL is defined as the Clearance of livmoniplimab.
CL of Budigalimab | Up to Approximately 3.5 Years
  CL is defined as the Clearance of budigalimab.
Volume of Distribution (Vd) of Livmoniplimab | Up to Approximately 3.5 Years
  Vd is defined as the volume of distribution of livmoniplimab.
Vd of Budigalimab | Up to Approximately 3.5 Years
  Vd is defined as the volume of distribution of budigalimab.
Incidence of Anti-Drug Antibodies (ADAs) of Livmoniplimab | Up to Approximately 3.5 Years
  Incidence of anti-drug antibodies of livmoniplimab.
ADAs of Budigalimab | Up to Approximately 3.5 Years
  Incidence of anti-drug antibodies of budigalimab.
Incidences of Neutralizing Anti-Drug Antibodies (nADAs) of Livmoniplimab | Up to Approximately 3.5 Years
  Incidences of neutralizing anti-drug antibodies of livmoniplimab.
Incidences of nADAs of Budigalimab | Up to Approximately 3.5 Years
  Incidences of neutralizing anti-drug antibodies of budigalimab.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (37):
- United States (11):
  - Highlands Oncology Group - Springdale /ID# 270290, Springdale, Arkansas
  - University of California San Francisco - Mission Bay /ID# 270289, San Francisco, California
  - Yale University School of Medicine /ID# 270449, New Haven, Connecticut
  - Medical Oncology Hematology Consultants /ID# 271347, Newark, Delaware
  - Florida Cancer Specialists - North /ID# 271215, St. Petersburg, Florida
  - Icahn School of Medicine at Mount Sinai /ID# 270272, New York, New York
  - University Hospitals Cleveland Medical Center /ID# 271010, Cleveland, Ohio
  - The Ohio State University /ID# 271349, Columbus, Ohio
  - SCRI Oncology Partners /ID# 270439, Nashville, Tennessee
  - Texas Oncology - Austin Central /ID# 271284, Austin, Texas
  - Utah Cancer Specialist /ID# 270810, Salt Lake City, Utah
- Centre Hospitalier Affilié Universitaire de Québec - Hôpital de l'Enfant-Jésus /ID# 271635, Québec, Quebec, Canada
- France (3):
  - Institut Paoli-Calmettes /ID# 270580, Marseille, Bouches-du-Rhone
  - Hôpital Foch /ID# 270573, Suresnes, Hauts-de-Seine
  - Institut Gustave Roussy /ID# 270575, Villejuif, Île-de-France Region
- Israel (5):
  - Meir Medical Center /ID# 270108, Kfar Saba, Central District
  - The Chaim Sheba Medical Center /ID# 270096, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 270106, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 270105, Haifa
  - Rabin Medical Center /ID# 270107, Petah Tikva
- Japan (4):
  - Hirosaki University Hospital /ID# 270531, Hirosaki, Aomori
  - Fukushima Medical University Hospital /ID# 270752, Fukushima, Fukushima
  - University of Tsukuba Hospital /ID# 270354, Tsukuba, Ibaraki
  - Kanazawa University Hospital /ID# 270473, Kanazawa, Ishikawa-ken
- Poland (2):
  - Aidport Sp. z o.o. /ID# 270049, Skórzewo, Greater Poland Voivodeship
  - Narodowy Instytut Onkologii Im. Marii Sklodowskiej-Curie Panstwowy Instytut Bada /ID# 270046, Warsaw, Masovian Voivodeship
- South Korea (5):
  - National Cancer Center /ID# 270453, Goyang-si, Gyeonggido
  - Chonnam National University Hwasun Hospital /ID# 271299, Hwasun-gun, Jeonranamdo
  - Yonsei University Health System Severance Hospital /ID# 270317, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 270898, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 270318, Seoul, Seoul Teugbyeolsi
- Spain (6):
  - Parc de Salut Mar - Hospital del Mar /ID# 270173, Barcelona
  - Hospital Universitario Vall d'Hebron /ID# 269783, Barcelona
  - Hospital Clinic de Barcelona /ID# 269789, Barcelona
  - Hospital MD Anderson Cancer Center Madrid /ID# 269780, Madrid
  - Hospital Clinico San Carlos /ID# 269786, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 269782, Seville

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-204